CLINICAL TRIAL: NCT05956756
Title: Effectiveness of Health and Resilience Programming for Occupational Therapy Students
Brief Title: Resilience Programming for Occupational Therapy Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5220395
Record Dates: First submitted 2023-07-12; First posted 2023-07-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Health and Wellbeing of Occupational Therapy Students
MeSH Terms: interventions — Health

STUDY DESIGN:
Intervention Model Description: This study will utilize a quasi-experimental design to explore the effectiveness of health and resilience programming for occupational therapy students while they are enrolled in the program. Pre and post data will be gathered through questionnaires. Additionally, qualitative data will be obtained from student discussion board posts/assignments, interviews or focus groups will be used to supplement the quantitative data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Occupational therapy students will engage in health and resiliency programming as part of their course work over their three year program.
  Interventions: Behavioral: Health and resiliency programming

INTERVENTIONS:
Behavioral: Health and resiliency programming — Students will engage in resilience programming as part of their regular coursework including mindfulness training, lifestyle medicine interventions, and creating a coping plan.

SUMMARY:
The purpose of this study is to explore the effectiveness of integrated health and resiliency programs into the Entry-Level Doctor of Occupational therapy curriculum.

The objectives are to:

1. Determine if students perceive health and resiliency programming as beneficial for their health and well-being
2. Determine if students' lifestyle behaviors, self-esteem, attachment security, and mindfulness improve with health and resiliency programming
3. Determine if students' symptoms of depression and anxiety reduce after participating in health and resiliency programs

Students will engage in resilience programming as part of their regular coursework and be invited to complete pre and post assessments to test the effectiveness of programming.

DETAILED DESCRIPTION:
University students are experiencing more challenges with anxiety, depression, and mental health. Health and resiliency programs embedded into the 3-year course curriculum may improve student health and wellness.

This study will utilize a quasi-experimental design to explore the effectiveness of health and resilience programming for occupational therapy students while they are enrolled in the program. Pre and post data will be gathered through questionnaires. Additionally, qualitative data will be obtained from student discussion board posts/assignments, interviews or focus groups will be used to supplement the quantitative data.

The purpose of this study is to explore the effectiveness of integrated health and resiliency programs into the Entry-Level Doctor of Occupational Therapy curriculum.

Objectives:

Determine if students perceive health and resiliency programming as beneficial for their health and well-being

Determine if students' lifestyle behaviors, self-esteem, attachment security, and mindfulness improve with health and resiliency programming

Determine if students' symptoms of depression and anxiety reduce after participating in health and resiliency programs

ELIGIBILITY:
Inclusion Criteria:

* students enrolled in the Entry Level Doctor of Occupational Therapy program at Loma Linda University
* Enrolled during June 2023 to June 2029
* Between 18-65 years of age
* Of any gender
* Of any ethnic background

Exclusion Criteria:

* N/A

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Health Promoting Lifestyle II (Walker, Sechrist, & Pender, 1987) | Three years
  This questionnaire contains 52 statements about respondents' present way of life or personal habits. Respondents are asked to respond to each item as accurately as possible on a 4-point Likert scale (never, sometimes, often, routinely). Example items include "Inspect my body at least monthly for physical changes/danger signs".
Rosenberg Self-Esteem Scale (Rosenberg, 1989) | Three years
  Include a list of 10 statements dealing with general feelings about oneself. Respondents are asked to indicate how strongly they agree or disagree with each statement on a 4-point Likert scale (strongly agree, agree, disagree, strongly disagree). An example item is "I am able to do things as well as most other people."
State Adult Attachment Measure (Gillath et al., 2009) | Three years
  Contains 21 statements concerning how the respondent feels right now in their relationship with others and self. Respondents indicate how much they agree or disagree with the statement as it reflects their current feelings on a 7-point sliding scale with 7 indicating 'agree strongly'. An example statement is "I wish someone close could see me now."
Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2001) | Three years
  Asks respondents to indicate how often they have been bothered by any of the following nine problems listed, over the last 2 weeks. Respondents use a 4-point Likert scale (not at all, several days, more than half the days, nearly everyday). An example statement is "Poor appetite or overeating."
General Anxiety Disorder (GAD-7; Williams, 2014) | Three years
  Asks respondents to indicate how often they have been bothered by any of the following seven problems listed, over the last 2 weeks. Respondents use a 4-point Likert scale (not at all, several days, more than half the days, nearly everyday). An example problem is "Not being able to stop or control worrying."
15-Facet mindfulness questionnaire (Baer et al., 2008) | Three years
  Contains 15-items related to mindfulness. Respondents rate how much they agree with each item on a 5-point Likert scale (very often or always, often true, sometimes true, rarely true, very rarely true). An example item is "When I have distressing thoughts or images I just notice them and let them go."

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda Universtiy, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No
We plan to share data from the overall group, reporting on averages, ranges and statistical output.